CLINICAL TRIAL: NCT02854332
Title: Evaluation of Repetitive Magnetic Stimulation Versus Direct Current Stimulation, in Chronic Neuropathic and Drug-resistant Pain Treatment
Brief Title: Analgesic Stimulation Non-invasive of the Motor Cortex
Acronym: DOLORIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 38RC14.130
Record Dates: First submitted 2016-07-25; First posted 2016-08-03 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-07

CONDITIONS: Neuropathic Chronic Pain
Keywords: Pain; Analgesic; Stimulation; Motor Cortex
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MRI by rTMS (Active Comparator): Patients which received an MRI study of cortical plasticity by rTMS.
  Interventions: Device: rTMS session
- MRI by tDCS (Active Comparator): Patients which received an MRI study of cortical plasticity by tDCS.
  Interventions: Device: tDCS session

INTERVENTIONS:
Device: tDCS session — Direct current transcranial magnetic stimulation
  Other Names: MRI
  Arms: MRI by tDCS
Device: rTMS session — Repetitive transcranial magnetic stimulation.
  Other Names: MRI
  Arms: MRI by rTMS

SUMMARY:
Prevalence of neuropathic pain raise to 6.9 % in the general population and can reach more than 58 % for patients that carry a lesion of the spinal cord. This pathological condition stays a major health problem, particularly as the efficacity of available treatments is currently limited. Only 30 to 40% of patients are relieved of more than 50% of their pain by a pharmacological approach.

In case of failure, drug treatments or in addition of these ones, stimulation of the motor cortex is a therapeutic path proposed by Tsubokawa since the beginning of 1990s, but that found its place for neuropathic drug-resistant pain management only since a decade. Neurophysiologic mechanisms of the analgesic efficacity of the motor cortex stimulation are still little understood. This stimulation can be realised in a chronic and invasive way with implanted electrodes. This process allow a lasting relief for about half of operated persons, without the possibility to identify clinical selection criterion reliable for potentially responding patients for this technique.

Recently, two electrophysiological non invasive techniques have been developed, allowing to get an analgesic stimulation of the motor cortex: the repetitive transcranial magnetic stimulation (rTMS) and the direct current transcranial magnetic stimulation (tDCS).

The main goal of this study is to compare the importance of analgesic effect of tDCS in chronic drug-resistant neurophysiologic pains to the one get thanks to a reference method of stimulation non invasive of the motor cortex, the rTMS whose analgesic effect is already validated by data of the literature.

ELIGIBILITY:
Inclusion Criteria:

* Persons affiliated to national social security.
* Patients that have given their signed free consent.
* Patients from 18 to 80 years, men or women, carriers of a chronic neuropathic pain (since more than a year ; EVN > 2during week S0) drug resistant, unilateral, involving at least the superior member and/or hemi-face, whose analgesic treatment is stable from at least one month.
* Patients whose drug resistance conduce their referent Algologist (specialist in pain medicine) to study the possibility to propose them alternative therapeutic solutions nonpharmacological and to start a pre-surgical examination.

Exclusion Criteria:

* History of drug addiction, migraine, epilepsy.
* Presence of ferromagnetic intracranial equipment or a stimulating implanted (pace-maker, stimulation of basal ganglia, vagus nerve stimulator).
* Introduction of a new analgesic treatment since at least a month.
* Pregnant, parturient or breastfeeding women. The absence of effective contraception during all the study for patients of childbearing age.
* Persons deprived of liberty by judicial or administrative decision, person under legal protection.
* Counter-argument to MRI.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
High-frequency | Half an hour
  rTMS session : repetitive transcranial magnetic stimulation.
  MRI
High-frequency | Half an hour
  tDCS session : direct current transcranial magnetic stimulation.
  MRI

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Hodaj, Doctor, Principal Investigator — Grenoble Hospital University
Locations (1):
- UniversityHospitalGrenoble, La Tronche, France

REFERENCES:
- [Background] Andre-Obadia N, Garcia-Larrea L, Garassus P, Mauguiere F. Timing and characteristics of perceptual attenuation by transcranial stimulation: a study using magnetic cortical stimulation and somatosensory-evoked potentials. Psychophysiology. 1999 Jul;36(4):476-83. doi: 10.1017/s0048577299971676. PMID 10432797
- [Background] Andre-Obadia N, Mertens P, Gueguen A, Peyron R, Garcia-Larrea L. Pain relief by rTMS: differential effect of current flow but no specific action on pain subtypes. Neurology. 2008 Sep 9;71(11):833-40. doi: 10.1212/01.wnl.0000325481.61471.f0. PMID 18779511
- [Background] Andre-Obadia N, Peyron R, Mertens P, Mauguiere F, Laurent B, Garcia-Larrea L. Transcranial magnetic stimulation for pain control. Double-blind study of different frequencies against placebo, and correlation with motor cortex stimulation efficacy. Clin Neurophysiol. 2006 Jul;117(7):1536-44. doi: 10.1016/j.clinph.2006.03.025. Epub 2006 Jun 5. PMID 16753335
- [Background] Attal N, Cruccu G, Haanpaa M, Hansson P, Jensen TS, Nurmikko T, Sampaio C, Sindrup S, Wiffen P; EFNS Task Force. EFNS guidelines on pharmacological treatment of neuropathic pain. Eur J Neurol. 2006 Nov;13(11):1153-69. doi: 10.1111/j.1468-1331.2006.01511.x. PMID 17038030
- [Background] Barker AT, Freeston IL, Jabinous R, Jarratt JA. Clinical evaluation of conduction time measurements in central motor pathways using magnetic stimulation of human brain. Lancet. 1986 Jun 7;1(8493):1325-6. doi: 10.1016/s0140-6736(86)91243-2. No abstract available. PMID 2872449
- [Background] Bouhassira D, Attal N, Fermanian J, Alchaar H, Gautron M, Masquelier E, Rostaing S, Lanteri-Minet M, Collin E, Grisart J, Boureau F. Development and validation of the Neuropathic Pain Symptom Inventory. Pain. 2004 Apr;108(3):248-257. doi: 10.1016/j.pain.2003.12.024. PMID 15030944
- [Background] Bouhassira D, Lanteri-Minet M, Attal N, Laurent B, Touboul C. Prevalence of chronic pain with neuropathic characteristics in the general population. Pain. 2008 Jun;136(3):380-387. doi: 10.1016/j.pain.2007.08.013. Epub 2007 Sep 20. PMID 17888574
- [Background] Cruccu G, Aziz TZ, Garcia-Larrea L, Hansson P, Jensen TS, Lefaucheur JP, Simpson BA, Taylor RS. EFNS guidelines on neurostimulation therapy for neuropathic pain. Eur J Neurol. 2007 Sep;14(9):952-70. doi: 10.1111/j.1468-1331.2007.01916.x. PMID 17718686
- [Background] Fregni F, Boggio PS, Lima MC, Ferreira MJ, Wagner T, Rigonatti SP, Castro AW, Souza DR, Riberto M, Freedman SD, Nitsche MA, Pascual-Leone A. A sham-controlled, phase II trial of transcranial direct current stimulation for the treatment of central pain in traumatic spinal cord injury. Pain. 2006 May;122(1-2):197-209. doi: 10.1016/j.pain.2006.02.023. Epub 2006 Mar 27. PMID 16564618
- [Background] Fregni F, Freedman S, Pascual-Leone A. Recent advances in the treatment of chronic pain with non-invasive brain stimulation techniques. Lancet Neurol. 2007 Feb;6(2):188-91. doi: 10.1016/S1474-4422(07)70032-7. PMID 17239806
- [Background] Fregni F, Gimenes R, Valle AC, Ferreira MJ, Rocha RR, Natalle L, Bravo R, Rigonatti SP, Freedman SD, Nitsche MA, Pascual-Leone A, Boggio PS. A randomized, sham-controlled, proof of principle study of transcranial direct current stimulation for the treatment of pain in fibromyalgia. Arthritis Rheum. 2006 Dec;54(12):3988-98. doi: 10.1002/art.22195. PMID 17133529
- [Background] Fregni F, Pascual-Leone A. Technology insight: noninvasive brain stimulation in neurology-perspectives on the therapeutic potential of rTMS and tDCS. Nat Clin Pract Neurol. 2007 Jul;3(7):383-93. doi: 10.1038/ncpneuro0530. PMID 17611487
- [Background] Garcia-Larrea L, Peyron R. Motor cortex stimulation for neuropathic pain: From phenomenology to mechanisms. Neuroimage. 2007;37 Suppl 1:S71-9. doi: 10.1016/j.neuroimage.2007.05.062. Epub 2007 Jun 29. PMID 17644413
- [Background] H. Hodaj, C. Maindet Dominici ,JP. Alibeu. Intérêt de la neuronavigation dans la pratique de la stimulation magnétique transcrânienne repetitive (SMTr) Douleurs, 2011, Vol.12 A77
- [Background] Hodaj H, Alibeu JP, Dominici C, D, Szekely D, Jacquot C. Traitement des douleurs réfractaires de la face par la stimulation magnétique transcranienne répétitive (SMTr) : étude ouverte sur une année Douleurs ; 2010, Vol. 11, 280-287
- [Background] Hodaj H, Pellat J, Szekely D, Alibeu JP, Bougerol T, Jacquot C. Utilisation de la stimulation magnétique transcranienne répétitive(SMTr) dans le traitement de la douleur neuropathique chronique résistante aux thérapeutiques conventionnelles. Douleurs, 2007,8, 1S62
- [Background] Khedr EM, Kotb H, Kamel NF, Ahmed MA, Sadek R, Rothwell JC. Longlasting antalgic effects of daily sessions of repetitive transcranial magnetic stimulation in central and peripheral neuropathic pain. J Neurol Neurosurg Psychiatry. 2005 Jun;76(6):833-8. doi: 10.1136/jnnp.2004.055806. PMID 15897507
- [Background] Lefaucheur JP, Drouot X, Menard-Lefaucheur I, Nguyen JP. Neuropathic pain controlled for more than a year by monthly sessions of repetitive transcranial magnetic stimulation of the motor cortex. Neurophysiol Clin. 2004 Apr;34(2):91-5. doi: 10.1016/j.neucli.2004.02.001. PMID 15130555
- [Background] Leo RJ, Latif T. Repetitive transcranial magnetic stimulation (rTMS) in experimentally induced and chronic neuropathic pain: a review. J Pain. 2007 Jun;8(6):453-9. doi: 10.1016/j.jpain.2007.01.009. Epub 2007 Apr 16. PMID 17434804
- [Background] McCann UD, Kimbrell TA, Morgan CM, Anderson T, Geraci M, Benson BE, Wassermann EM, Willis MW, Post RM. Repetitive transcranial magnetic stimulation for posttraumatic stress disorder. Arch Gen Psychiatry. 1998 Mar;55(3):276-9. doi: 10.1001/archpsyc.55.3.276. No abstract available. PMID 9510224
- [Background] Mertens P, Nuti C, Sindou M, Guenot M, Peyron R, Garcia-Larrea L, Laurent B. Precentral cortex stimulation for the treatment of central neuropathic pain: results of a prospective study in a 20-patient series. Stereotact Funct Neurosurg. 1999;73(1-4):122-5. doi: 10.1159/000029769. PMID 10853116
- [Background] Merzagora AC, Foffani G, Panyavin I, Mordillo-Mateos L, Aguilar J, Onaral B, Oliviero A. Prefrontal hemodynamic changes produced by anodal direct current stimulation. Neuroimage. 2010 Feb 1;49(3):2304-10. doi: 10.1016/j.neuroimage.2009.10.044. Epub 2009 Oct 21. PMID 19853048
- [Background] Migita K, Uozumi T, Arita K, Monden S. Transcranial magnetic coil stimulation of motor cortex in patients with central pain. Neurosurgery. 1995 May;36(5):1037-9; discussion 1039-40. doi: 10.1227/00006123-199505000-00025. PMID 7540735
- [Background] Nguyen JP, Lefaucheur JP, Decq P, Uchiyama T, Carpentier A, Fontaine D, Brugieres P, Pollin B, Feve A, Rostaing S, Cesaro P, Keravel Y. Chronic motor cortex stimulation in the treatment of central and neuropathic pain. Correlations between clinical, electrophysiological and anatomical data. Pain. 1999 Sep;82(3):245-251. doi: 10.1016/S0304-3959(99)00062-7. PMID 10488675
- [Background] Nitsche MA, Fricke K, Henschke U, Schlitterlau A, Liebetanz D, Lang N, Henning S, Tergau F, Paulus W. Pharmacological modulation of cortical excitability shifts induced by transcranial direct current stimulation in humans. J Physiol. 2003 Nov 15;553(Pt 1):293-301. doi: 10.1113/jphysiol.2003.049916. Epub 2003 Aug 29. PMID 12949224
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] Nuti C, Peyron R, Garcia-Larrea L, Brunon J, Laurent B, Sindou M, Mertens P. Motor cortex stimulation for refractory neuropathic pain: four year outcome and predictors of efficacy. Pain. 2005 Nov;118(1-2):43-52. doi: 10.1016/j.pain.2005.07.020. Epub 2005 Oct 7. PMID 16214292
- [Background] O'Connell NE, Wand BM, Marston L, Spencer S, Desouza LH. Non-invasive brain stimulation techniques for chronic pain. A report of a Cochrane systematic review and meta-analysis. Eur J Phys Rehabil Med. 2011 Jun;47(2):309-26. Epub 2011 Apr 14. PMID 21494222
- [Background] Pascual-Leone A, Catala MD, Pascual-Leone Pascual A. Lateralized effect of rapid-rate transcranial magnetic stimulation of the prefrontal cortex on mood. Neurology. 1996 Feb;46(2):499-502. doi: 10.1212/wnl.46.2.499. PMID 8614521
- [Background] Paulus W. Transcranial direct current stimulation (tDCS). Suppl Clin Neurophysiol. 2003;56:249-54. doi: 10.1016/s1567-424x(09)70229-6. PMID 14677402
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Rossini PM, Barker AT, Berardelli A, Caramia MD, Caruso G, Cracco RQ, Dimitrijevic MR, Hallett M, Katayama Y, Lucking CH, et al. Non-invasive electrical and magnetic stimulation of the brain, spinal cord and roots: basic principles and procedures for routine clinical application. Report of an IFCN committee. Electroencephalogr Clin Neurophysiol. 1994 Aug;91(2):79-92. doi: 10.1016/0013-4694(94)90029-9. No abstract available. PMID 7519144
- [Background] Stagg CJ, O'Shea J, Kincses ZT, Woolrich M, Matthews PM, Johansen-Berg H. Modulation of movement-associated cortical activation by transcranial direct current stimulation. Eur J Neurosci. 2009 Oct;30(7):1412-23. doi: 10.1111/j.1460-9568.2009.06937.x. Epub 2009 Sep 29. PMID 19788568
- [Background] Torrance N, Smith BH, Bennett MI, Lee AJ. The epidemiology of chronic pain of predominantly neuropathic origin. Results from a general population survey. J Pain. 2006 Apr;7(4):281-9. doi: 10.1016/j.jpain.2005.11.008. PMID 16618472
- [Background] Tsubokawa T, Katayama Y, Yamamoto T, Hirayama T, Koyama S. Chronic motor cortex stimulation in patients with thalamic pain. J Neurosurg. 1993 Mar;78(3):393-401. doi: 10.3171/jns.1993.78.3.0393. PMID 8433140
- [Background] Zaghi S, Thiele B, Pimentel D, Pimentel T, Fregni F. Assessment and treatment of pain with non-invasive cortical stimulation. Restor Neurol Neurosci. 2011;29(6):439-51. doi: 10.3233/RNN-2011-0615. PMID 22124038